CLINICAL TRIAL: NCT00383305
Title: Brain-Cooling for the Treatment of Perinatal Hypoxic-Ischemic Encephalopathy
Brief Title: CoolCap Trial, Treatment of Perinatal Hypoxic-Ischemic Encephalopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Olympic Medical (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IDE G990037; PMA P040025; HIE-0198
Record Dates: First submitted 2006-09-29; First posted 2006-10-03 (Estimated); Last update posted 2006-10-03 (Estimated); Status verified 2006-09

CONDITIONS: Neonatal Hypoxic-Ischemic Encephalopathy (HIE)
Keywords: neonatal; hypoxic; ischemic; encephalopathy; HIE; birth asphyxia; neonatal encephalopathy; Asphyxia Neonatorum; hypothermia, therapeutic; brain cooling; selective head cooling
MeSH Terms: conditions — Hypoxia; Ischemia; Brain Diseases; Asphyxia Neonatorum; Hypothermia

INTERVENTIONS:
Device: Cool-Cap

SUMMARY:
This is a research study of head cooling. Its goal is to determine whether cooling babies' heads can reduce or prevent brain damage that may have resulted from temporarily reduced oxygen supply to the brain. In this study, half of the babies (selected at random) will have a special cooling cap with circulating water placed on their head for 72 hours to lower the temperature of their brain. The rest of the baby's body will be maintained at a defined temperature by a standard overhead radiant heater. The study protocol includes the taking and analysis of blood samples, performance of brain wave tests, imaging of the brain by ultrasound, and other tests as clinically indicated. Neurodevelopmental outcome will also be assessed at 18 months of age.

DETAILED DESCRIPTION:
The objective of this study is to determine whether head cooling with mild systemic hypothermia in term infants following perinatal asphyxia is a safe procedure that improves survival without neurodevelopmental disability. Outcome will be assessed by survival and neurological and neurodevelopmental testing at 18 months of age.

Within 6 hours of birth, infants will be randomized to either a non-cooled control group with rectal temperature kept at 37+/-0.5 degC or to head cooling with mild systemic hypothermia as follows. A cooling device capable of circulating cool water in a temperature-regulated manner through a cap fitted around the infant's scalp will cool the head. The core rectal temperature of the infant will be maintained at 34.5+/-0.5 degC by adjusting the cap water temperature. The infant's rectal, nasopharyngeal, scalp (fontanel), and skin (abdominal) temperatures will be continuously monitored. Also, metabolic, cardiovascular, pulmonary and coagulation laboratory measurements will be assessed at predefined time points. Cooling will be maintained for 72 hours, followed by four hours of rewarming, with the goal of raising the rectal temperature to normal body temperature by 0.5 degC per hour. The outcome measure of severe neurodevelopmental disability and survival rates at 18 months of age will be assessed by blinded, independent observers.

ELIGIBILITY:
Inclusion Criteria:

Infants are assessed sequentially by criteria A, B and C listed below. Infant must meet all three criteria to be eligible for trial enrollment.

* Criteria A: Infants >= 36 weeks gestation admitted to the NICU with ONE of the following:

  * Apgar score of <= 5 at 10 minutes after birth;
  * Continued need for resuscitation, including endotracheal or mask ventilation, at 10 minutes after birth;
  * Acidosis defined as either umbilical cord pH or any arterial pH within 60 minutes of birth < 7.00; or
  * Base Deficit <= -16 mmol/L in umbilical cord blood sample OR any blood sample within 60 minutes of birth (arterial or venous blood).
* Criteria B: Moderate to severe encephalopathy consisting of altered state of consciousness (as shown by lethargy, stupor, or coma) AND at least one or more of the following:

  * Hypotonia;
  * Abnormal reflexes, including oculomotor or pupillary abnormalities;
  * An absent or weak suck;
  * Clinical seizures
* Criteria C: At least 20 minutes duration of amplitude integrated EEG (aEEG/CFM) recording that shows abnormal background aEEG/CFM activity or seizures. The aEEG/CFM is to be performed from one hour of age. If subsequently an abnormal aEEG/CFM is recorded before 5.5 hours of age, the infant is then eligible for enrollment. The aEEG is not to be performed within 30 minutes of IV anticonvulsant therapy as this may cause suppression of EEG activity. In particular, high dose prophylactic anticonvulsant therapy (e.g., >20 mg/kg phenobarbitone) is not to be given prior to performing the aEEG/CFM.

Exclusion Criteria:

* Infant expected to be > 5.5 hours of age at the time of randomization
* Prophylactic administration of high dose anticonvulsants (e.g., >20 mg/kg phenobarbitone). After trial entry phenobarbitone or other anticonvulsant therapy is allowed to be given as clinically indicated to treat seizures.
* Major congenital abnormalities, such as diaphragmatic hernia requiring ventilation, or congenital abnormalities suggestive of chromosomal anomaly or other syndromes that include brain dysgenesis
* Imperforate anus
* Evidence of head trauma or skull fracture causing major intracranial hemorrhage
* Infant < 1,800 g birth weight
* Head circumference < (mean - 2SD) for gestation if birth weight and length are > (mean - 2SD)
* Infant "in extremis" (i.e. an infant for whom no other additional intensive management would be offered in the judgment of the attending neonatologist)
* Unavailability of essential equipment (e.g., Cool-Cap, aEEG/CFM)
* Planned concurrent participation in other experimental treatments

Ages: 1 Hour to 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 235
Dates: Start 1999-07; Study Completion 2003-09

PRIMARY OUTCOMES:
Combined death or severe neurodevelopmental disability in the first 18 months of life.

SECONDARY OUTCOMES:
Length of hospitalization during NICU course in those surviving to discharge and for whom support was not withdrawn.
Multi-organ dysfunction (3 or more organ systems) in the neonatal period.
Rate of multiple handicap in survivors (Multiple handicap will be defined as the presence of any two of the following in an infant: neuromotor disability (Level 3-5 on GMF classification), mental delay, epilepsy, cortical visual impairment, sensorineural
Bayley PDI score
Sensorineural hearing loss >= 40 dB
Epilepsy: recurrent seizures beyond the neonatal period, requiring anticonvulsant therapy at the time of assessment.
Microcephaly: head circumference < (mean - 2SD)

CONTACTS AND LOCATIONS:
Overall Officials: Peter D Gluckman, M.D., Principal Investigator — The Liggins Institute, University of Auckland; Auckland, New Zealand; John S. Wyatt, M.D., Principal Investigator — University College London; London, UK; Alistair J Gunn, M.D., Ph.D., Study Director — Department of Physiology, University of Auckland; Auckland, New Zealand
Locations (27):
- United States (19):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - University of California San Diego Medical Center (Hillcrest), San Diego, California
  - University of California San Francisco Children's Hospital, San Francisco, California
  - Children's Hospital of Denver, Denver, Colorado
  - Children's Memorial Hospital / Prentice Women's Hospital, Chicago, Illinois
  - University of Illinois at Chicago Medical Center, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan Medical Center - Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital and Clinics of Minneapolis, Minneapolis, Minnesota
  - Schneider Children's Hospital, New Hyde Park, New York
  - Children's Hospital of new York - Presbyterian (Columbia University), New York, New York
  - Golisano Children's Hospital at Strong, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Children's Hospital of Oklahoma, Oklahoma City, Oklahoma
  - AI Dupont Children's Hospital at Thomas Jefferson University Medical Center, Philadelphia, Pennsylvania
  - Magee Women's Hospital / Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Canada (3):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Children's Hospital of Eastern Ontario / The Ottawa Hospital, Ottawa, Ontario
- University of Auckland - National Women's Hospital, Auckland, New Zealand
- United Kingdom (4):
  - Southmead Hospital, Bristol, England
  - St. Michael's Hospital, Bristol
  - Hammersmith Hospital, London
  - University College Hospital, London

REFERENCES:
- [Result] Gluckman PD, Wyatt JS, Azzopardi D, Ballard R, Edwards AD, Ferriero DM, Polin RA, Robertson CM, Thoresen M, Whitelaw A, Gunn AJ. Selective head cooling with mild systemic hypothermia after neonatal encephalopathy: multicentre randomised trial. Lancet. 2005 Feb 19-25;365(9460):663-70. doi: 10.1016/S0140-6736(05)17946-X. PMID 15721471
- [Result] Dutta S, Pradeep GC, Narang A. Selective head cooling after neonatal encephalopathy. Lancet. 2005 May 7-13;365(9471):1619; author reply 1619-20. doi: 10.1016/S0140-6736(05)66503-8. No abstract available. PMID 15885292
- [Result] Bello SO. Selective head cooling after neonatal encephalopathy. Lancet. 2005 May 7-13;365(9471):1619; author reply 1619-20. doi: 10.1016/S0140-6736(05)66504-X. No abstract available. PMID 15885291
- [Result] Rutherford MA, Azzopardi D, Whitelaw A, Cowan F, Renowden S, Edwards AD, Thoresen M. Mild hypothermia and the distribution of cerebral lesions in neonates with hypoxic-ischemic encephalopathy. Pediatrics. 2005 Oct;116(4):1001-6. doi: 10.1542/peds.2005-0328. PMID 16199715
- [Derived] Basu SK, Salemi JL, Gunn AJ, Kaiser JR; CoolCap Study Group. Hyperglycaemia in infants with hypoxic-ischaemic encephalopathy is associated with improved outcomes after therapeutic hypothermia: a post hoc analysis of the CoolCap Study. Arch Dis Child Fetal Neonatal Ed. 2017 Jul;102(4):F299-F306. doi: 10.1136/archdischild-2016-311385. Epub 2016 Oct 31. PMID 27799322
- [Derived] Basu SK, Kaiser JR, Guffey D, Minard CG, Guillet R, Gunn AJ; CoolCap Study Group. Hypoglycaemia and hyperglycaemia are associated with unfavourable outcome in infants with hypoxic ischaemic encephalopathy: a post hoc analysis of the CoolCap Study. Arch Dis Child Fetal Neonatal Ed. 2016 Mar;101(2):F149-55. doi: 10.1136/archdischild-2015-308733. Epub 2015 Aug 17. PMID 26283669